CLINICAL TRIAL: NCT02491437
Title: A Randomized, Open-label, Two-arm, Multicenter Study Comparing the Efficacy, Safety and Tolerability of Oral Dydrogesterone 30 mg Daily Versus Crinone 8% Intravaginal Progesterone Gel 90 mg Daily for Luteal Support in In-Vitro Fertilization (LOTUS II)
Brief Title: A Study Comparing the Efficacy, Safety and Tolerability of Oral Dydrogesterone 30 mg Daily Versus Crinone 8% Intravaginal Progesterone Gel 90 mg Daily for Luteal Support in In-Vitro Fertilization (LOTUS II)
Acronym: LOTUS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: PRA Health Sciences (Industry); Datamap (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-625; 2012-002993-29 (EudraCT Number)
Record Dates: First submitted 2015-06-16; First posted 2015-07-08 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Dydrogesterone; Crinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dydrogesterone tablets 3x10 mg (Experimental): Dydrogesterone tablets 3x10 mg
  Interventions: Drug: Dydrogesterone 30 mg
- Crinone 8% intravaginal progesterone gel 90 mg (Experimental): Crinone 8% intravaginal progesterone gel 90 mg
  Interventions: Drug: intravaginal progesterone gel 90 mg

INTERVENTIONS:
Drug: Dydrogesterone 30 mg — Oral Dydrogesterone 10 mg tablets tid
  Arms: Dydrogesterone tablets 3x10 mg
Drug: intravaginal progesterone gel 90 mg
  Other Names: Crinone 8% intravaginal progesterone gel 90 mg
  Arms: Crinone 8% intravaginal progesterone gel 90 mg

SUMMARY:
The purpose of this randomized, two-arm and open label study is to demonstrate that the treatment of a daily dose of 3x10mg dydrogesterone orally is as effective and safe as the daily dose Crinone 8% intravaginal progesterone gel 90 mg for the luteal support in women who are unable to conceive a child and are undergoing IVF. The treatment will start on the day of oocyte retrieval and continue until pregnancy is negative or until week 12 gestation.

Patients will be followed during treatment until 30 days after delivery to record any safety and tolerability data of the patient and their newborn (s).

DETAILED DESCRIPTION:
"This article has been accepted for publication in Human Reproduction published by Oxford University Press."

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Premenopausal females, age > 18 years < 42 years
* Non-smokers. For females who were past smokers, they must have stopped tobacco usage for at least 3 months prior screening visit
* Early follicular phase (Day 2-4) Follicle stimulating hormone (FSH) less than or equal to 15 IU/L and estradiol (E2)within normal limits at screening
* luteinizing hormone (LH), prolactin (PRL), T (testosterone) and thyroid-stimulating hormone (TSH), within the normal limits for the clinical laboratory, or considered not clinically significant by the Investigator within 6 months prior or at screening
* Documented history of infertility (e.g., unable to conceive for at least one year or for 6 months for women ≥ 38 years of age or bilateral tubal occlusion or absence)
* Normal transvaginal ultrasound at screening (or within 14 days prior of screening) without evidence of clinically significant abnormality consistent with finding adequate for Assisted Reproductive Technology (ART) with respect to uterus and adnexa (no hydrosalpinx or clinically relevant uterine fibroids)
* Subject is not pregnant , confirmed by negative pregnancy or by Investigator Judgement
* Clinically indicated protocol for induction of IVF with a fresh embryo
* Single or dual embryo transfer
* BMI ≥ 18 and ≤ 30 kg/m2

Exclusion Criteria:

* Evidence of cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatologic/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurologic/psychiatric, allergy, recent major surgery (< 3 months), or other relevant diseases as revealed by history, physical examination and/or laboratory assessments which could limit participation in or completion of the study;
* Acute urogenital disease
* Known allergic reactions to progesterone products
* Known allergic reactions to peanuts and peanut oil
* Intake of àny experimental drug or any participation in any other clinical trial within 30 days prior to study start
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subjects to participate in or to complete the study
* Current or recent substance abuse, including alcohol and tobacco (Note: Patients who stopped tobacco usage at least 3 months prior to screening visit would be allowed)
* History of chemotherapy or radiotherapy
* Patients with more than 3 unsuccessful IVF attempts
* Contraindication for pregnancy
* Refusal or inability to comply with the requirements of the study protocol for any reason, including scheduled clinic visits and laboratory tests
* History of recurrent pregnancy loss defined as 3 or more spontaneous miscarriages Acute urogenital disease

Ages: 19 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1034 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shreyansh Shah, MD, Study Director — Abbott
Locations (40):
- Australia (2):
  - Melbourne IVF, East Melbourne
  - IVF Australia - St George Private HospitalIVF Australia - St George Private Hospital, Kogarah
- Belgium (4):
  - Univerité Catholique de Louvain, Cliniques universitaires Saint-Luc, Brussels
  - Algemeen Ziekenhuis Jan Palfijn Gent, Ghent
  - UZ Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
- China (9):
  - Peking University People's Hospital, Beijing
  - Reproductive & Genetic Hospital of Citic -Xiangya, Changsha
  - West China Second University Hospital, Chengdu
  - Sun Yat-Sen Memorial Hsopiatl, Sun Yat-Sen University, Guangzhou
  - The Sixth Hospital of Sun Yat-Sen University, Guangzhou
  - The First Affiliate Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Germany (4):
  - Fertility Center Berlin, Berlin
  - Bielefeld Fertility Center, Bielefeld
  - Kinderwunschzentrum Dortmund, Dortmund
  - Universitäres Kinderwunschzentrum Lübeck, Lübeck
- Queen Mary Hospital, Hong Kong, Hong Kong
- India (9):
  - United CIIGMA Hospital, Aurangabad
  - MILANN (Bangalore Assisted Conception Center), Bangalore
  - Apollo Hospitals - Bangalore, Bangalore
  - All India Institute of Medical Sciences, Delhi
  - Max Hospital, Delhi
  - Institute of Reproductive Medicine, Kolkata
  - Ajanta Research Center, Ajanta Hospital and IVF center, Lucknow
  - Inamdar Multispecialty Hospital, Pune
  - Shree Hospital and Diagnostic Centre, Pune
- Russia (4):
  - Scientific Research Center of Obstetrics, Gynecology and Perinatology n. a. Ac. V. I. Kulakova, Moscow
  - CJSC "Nasledniki", Moscow
  - Saint-Petersburg State Budgetary Healtcare Institution "Maternity Hospital # 17", Saint Petersburg
  - CJSC "Center of Family Medicine", Yekaterinburg
- Singapore General Hospital, Singapore, Singapore
- Thailand (2):
  - Songklanagarind Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Ukraine (4):
  - Medical Centre of Infertility Treatment "Clinic of Professor Yuzko", Chernivtsi
  - "NADIYA" Clinic, Kiev
  - The Institute for Reproductive Medicine in Ukraine, Kiev
  - "Mother and Child" clinic, Kiev

REFERENCES:
- [Derived] Griesinger G, Blockeel C, Sukhikh GT, Patki A, Dhorepatil B, Yang DZ, Chen ZJ, Kahler E, Pexman-Fieth C, Tournaye H. Oral dydrogesterone versus intravaginal micronized progesterone gel for luteal phase support in IVF: a randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2212-2221. doi: 10.1093/humrep/dey306. PMID 30304457

RESULTS

PARTICIPANT FLOW:
Groups:
- Crinone 8% Intravaginal Progesterone Gel 90 mg: Crinone 8% intravaginal progesterone gel 90 mg
  intravaginal progesterone gel 90 mg OD
Period: Overall Study
Arm/Group | Dydrogesterone Tablets 3x10 mg | Crinone 8% Intravaginal Progesterone Gel 90 mg
Started | 520 | 514
Safety Sample | 518 | 512
Full Analysis Sample | 494 | 489
Completed | 168 | 157
Not Completed | 352 | 357

BASELINE CHARACTERISTICS:
Population: This is the full analysis sample
Groups:
- Total: Total of all reporting groups
Arm/Group | Dydrogesterone Tablets 3x10 mg | Crinone 8% Intravaginal Progesterone Gel 90 mg | Total
Number analyzed (Participants) | 494 | 489 | 983
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 494 | 489 | 983
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (4.4) | 31.6 (4.6) | 31.7 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 489 | 983
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 250 | 237 | 487
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 237 | 247 | 484
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 10 | 9 | 19
  Belgium | 80 | 85 | 165
  Hong Kong | 9 | 7 | 16
  China | 114 | 108 | 122
  Ukraine | 45 | 46 | 91
  Thailand | 13 | 12 | 25
  Australia | 3 | 2 | 5
  Germany | 78 | 79 | 157
  India | 103 | 100 | 203
  Russia | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Presence of Fetal Heart Beats at 12 Week's Gestation Determined by Transvaginal Ultrasound
Description: Pregnancy rate defined as the presence of fetal heart beats at 12 weeks' gestation determined by transvaginal ultrasound.
Time Frame: 12 weeks´ gestation
Population: Full Analysis Sample (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dydrogesterone Tablets 3x10 mg | Crinone 8% Intravaginal Progesterone Gel 90 mg
Number analyzed (Participants) | 494 | 489
percentage of participants | 38.7 [34.4 to 43.1] | 35.0 [30.7 to 39.4]

2. Secondary Outcome: Positive Pregnancy Test Rate (Percentage of Participants With a Positive Biochemical Pregnancy Test on Day 14 After Embryo Transfer)
Description: Positive biochemical pregnancy test on Day 14 after embryo transfer
Time Frame: Day 14 after embryo transfer
Population: Full Analysis Sample (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dydrogesterone Tablets 3x10 mg | Crinone 8% Intravaginal Progesterone Gel 90 mg
Number analyzed (Participants) | 494 | 489
percentage of participants | 47.4 [42.9 to 51.9] | 43.8 [39.3 to 48.3]

3. Secondary Outcome: Rate of Successful Completion of Pregnancy (Percentage of Participants With a Live Birth)
Description: Live birth rate (percentage of participants with a live birth)
Time Frame: After delivery (about 9 months after IVF)
Population: Full Analysis Sample (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dydrogesterone Tablets 3x10 mg | Crinone 8% Intravaginal Progesterone Gel 90 mg
Number analyzed (Participants) | 494 | 489
percentage of participants | 34.4 [30.2 to 38.8] | 32.5 [28.4 to 36.9]

4. Secondary Outcome: Physical Examination Newborn (Number of Delivered Newborns That Are Male or Female)
Description: The gender (number of delivered newborns that are male or female)
Time Frame: After delivery (about 9 months after IVF)
Population: Full Analysis Sample (FAS). These are the number of delivered babies from the mothers in the FAS
Measure: Number; unit: number of newborns
Arm/Group | Dydrogesterone Tablets 3x10 mg | Crinone 8% Intravaginal Progesterone Gel 90 mg
Number analyzed (Participants) | 205 | 188
number of newborns
  Gender male | 105 | 95
  Gender female | 100 | 93

ADVERSE EVENTS:
Time Frame: After signing of informed consent form until 30 days after birth, up to 11 months
Description: For Adverse Events reporting the safety sample was used consisting of all subjects which have received at least one administration of study drug (518 subjects in Dydrogesterone, 512 subjects in Micronized Progesterone)
Groups:
- Dydrogesterone Tablets 3x10 mg (Maternal): Dydrogesterone tablets 3x10 mg
  Dydrogesterone 30 mg: Oral Dydrogesterone 10 mg tablets tid
- Crinone 8% Intravaginal Progesterone Gel 90 mg (Maternal): Crinone 8% intravaginal progesterone gel 90 mg
  Intravaginal progesterone gel 90 mg OD
- Dydrogesterone Tablets (Fetus/Newborn): Maternal dosing of Dydrogesterone tablets 3x10 mg
  221 subjects at risk=205 live births + 16 abortions/stillbirths
- Crinone 8% Intravaginal Progesterone Gel (Fetus/Newborn): Maternal dosing of Crinone 8% intravaginal progesterone gel 90 mg
  201 subjects at risk = 188 live births + 13 abortions/stillbirths
Arm/Group | Dydrogesterone Tablets 3x10 mg (Maternal) | Crinone 8% Intravaginal Progesterone Gel 90 mg (Maternal) | Dydrogesterone Tablets (Fetus/Newborn) | Crinone 8% Intravaginal Progesterone Gel (Fetus/Newborn)
All-Cause Mortality (participants affected / at risk) | 0/518 | 0/512 | 4/221 | 0/201
Serious Adverse Events (participants affected / at risk) | 71/518 | 67/512 | 28/221 | 23/201
Other Adverse Events (participants affected / at risk) | 50/518 | 35/512 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dydrogesterone Tablets 3x10 mg (Maternal) (N=518) | Crinone 8% Intravaginal Progesterone Gel 90 mg (Maternal) (N=512) | Dydrogesterone Tablets (Fetus/Newborn) (N=221) | Crinone 8% Intravaginal Progesterone Gel (Fetus/Newborn) (N=201)
abortions spontaneous (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 14 (14) | 0 (0) | 0 (0)
maternal complications of pregnancy (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 11 (11) | 0 (0) | 0 (0)
labour onset and length abnormalities (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 12 (13) | 6 (7) | 0 (0) | 0 (0)
abortion not specified as induced or spontaneous (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 4 (4) | 0 (0) | 0 (0)
gestational age and weight conditions (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 6 (6) | 0 (0) | 0 (0)
still birth and foetal death (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Hypertension associated disorders of pregnancy (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
placental abnormalities (excl neoplasms) (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
haeomorrhagic complications of pregnancy (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
abortion related conditions and complications (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
pregnancy complicated by maternal disorders (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
amniotic fluid and cavity disorders of pregnancy (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
maternal complications of delivery (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
postpartum complications (related to the mother) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ovarium and fallopian tube disorders (related to the mother) (Reproductive system and breast disorders) | 11 (12) | 15 (15) | 0 (0) | 0 (0)
vulvovaginal disorders (related to the mother) (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Uterine disorders (related to the mother) (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
induced abortions (related to the mother) (Surgical and medical procedures) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
obstetric therapeutic procedures (related to the mother) (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
gastrointestinal and abdominal pains (excl oral and throat) (related to the mother) (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
flatulence, bloating and distension (related to the mother) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
large intestinal stenosis and obstruction (related to the mother) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
upper respiratory tract infections (related to the mother) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
urinary tract infections (related to the mother) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
viral infections (related to the mother) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
central nervous system vascular disorders (related to the mother) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
facial cranial nerve disorders (related to the mother) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
renal obstructive disorders (related to the mother) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
urinary tract signs and symptoms (related to the mother) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
non-site specific injuries (related to the mother) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
thyroid neoplasms malignant (related to the mother) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
peripheral embolism and thrombosis (related to the mother) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cardiac septal defects congenital (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 5 (5) | 7 (7)
cardiac disorders congenital NEC (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
persistant foetal circulation disorders (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
muskuloskeletal and connective tissue disorders of limbs congenital (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
renal disorders congenital (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
central nervous system disorder congenital NEC (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
great vessel disorders congenital (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
intestinal disorders congenital (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lymphatic system disorders congenital (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-site specific muscle disorders congenital (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sex chromosomal abnormalities (fetus/newborn) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lower respiratory tract and lung infections (fetus/newborn) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
sepsis, bacteraemia, viraemia and fungaemia NEC (fetus/newborn) (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
infections NEC (fetus/newborn) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
respiratory syncytial viral infections (fetus/newborn) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gestational age and weight conditions (fetus/newborn) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
foetal complications NEC (fetus/newborn) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
foetal growth complications (fetus/newborn) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
neonatal hypoxic conditions (fetus/newborn) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (6)
pulmonary oedemas (fetus/newborn) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
breathing abnormalities (fetus/newborn) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
respiratory failures (excl neonatal) (fetus/newborn) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
rate and rythm disorders NEC (fetus/newborn) (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
ischaemic coronary artery disorders (fetus/newborn) (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
encephalopathies NEC (fetus/newborn) (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
structural brain disorders NEC (fetus/newborn) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
hydrocephalic conditions (fetus/newborn) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
foetal and neonatal diagnostic procedures (fetus/newborn) (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
coagulopathies (fetus/newborn) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The number of fetus/newborn was 221 in the dydrogesterone group and 201 in the micronized progesterone group. Frequencies in the Adverse Event table are provided based on the safety sample.
colitis (excl infective) (fetus/newborn) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
intestinal ulcers and perforation NEC (fetus/newborn) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dydrogesterone Tablets 3x10 mg (Maternal) (N=518) | Crinone 8% Intravaginal Progesterone Gel 90 mg (Maternal) (N=512) | Dydrogesterone Tablets (Fetus/Newborn) (N=0) | Crinone 8% Intravaginal Progesterone Gel (Fetus/Newborn) (N=0)
Vaginal haemorrhage (Pregnancy, puerperium and perinatal conditions) | 50 (50) | 35 (35) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials, and allow sponsor sixty (60) days to review and comment on them.

If the Sponsor requests, the Site shall remove any Confidential Information (other than Study results) prior to submitting or presenting the materials.

DOCUMENTS (2):
  • Study Protocol (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT02491437/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT02491437/SAP_001.pdf